CLINICAL TRIAL: NCT01189253
Title: TRUSTS: A Phase IIB/III Multicenter Study Comparing the Efficacy of TRabectedin Administered as a 3-Hour or 24-Hour Infusion to Doxorubicin in Patients With Advanced or Metastatic Untreated Soft Tissue Sarcoma
Brief Title: Doxorubicin Hydrochloride or Trabectedin in Treating Patients With Previously Untreated Advanced or Metastatic Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Results of step1: none of the experimental arms fulfills expectations and the study will not continue as a phase III.
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-62091; EORTC-62091; 2009-014889-26 (EudraCT Number); EU-21059; PMAR-EORTC-62091; SARC-020
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Sarcoma
Keywords: stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; adult alveolar soft-part sarcoma; adult angiosarcoma; adult desmoplastic small round cell tumor; adult epithelioid sarcoma; adult extraskeletal chondrosarcoma; adult extraskeletal osteosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult malignant mesenchymoma; adult neurofibrosarcoma; adult synovial sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Alveolar Soft Part; Hemangiosarcoma; Desmoplastic Small Round Cell Tumor; Chondrosarcoma, Extraskeletal Myxoid; Fibrosarcoma; Leiomyosarcoma; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Neurofibrosarcoma; Sarcoma, Synovial | interventions — Doxorubicin; Trabectedin

ARMS (3):
- Doxorubicin 75 mg/m² every 3 weeks (Active Comparator): Doxorubicin administered on day 1 every 3 weeks for a maximum of 6 cycles
  Interventions: Drug: doxorubicin hydrochloride; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment
- Trabectedin IV 3 hours (Experimental): Trabectedin administered on day 1 every 3 weeks at the dose of 1.3 mg/m² until progression
  Interventions: Drug: trabectedin; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment
- Trabectedin IV 24 hours every 3 weeks (Experimental): Trabectedin administered on day 1 every 3 weeks at the dose of 1.5 mg/m² over 24 hours until progression
  Interventions: Drug: trabectedin; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: doxorubicin hydrochloride
  Arms: Doxorubicin 75 mg/m² every 3 weeks
Drug: trabectedin
  Arms: Trabectedin IV 24 hours every 3 weeks; Trabectedin IV 3 hours
Other: laboratory biomarker analysis
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride and trabectedin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether trabectedin is more effective than doxorubicin hydrochloride in treating patients with advanced or metastatic soft tissue sarcoma.

PURPOSE: This randomized phase II/III trial is studying the safety of trabectedin compared with doxorubicin hydrochloride and to see how well they work in treating patients with advanced or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate whether trabectedin given as first-line chemotherapy for patients with previously untreated advanced or metastatic malignant soft tissue sarcoma prolongs progression-free survival as compared to doxorubicin hydrochloride.
* To identify and validate biomarkers (including, but not limited to, XPG, BRCA1, RAD51, BRCA2, ATM and CHK1) of sensitivity to trabectedin in order to allow the selection of patients that benefit most from trabectedin treatment. (Optional translational research)

OUTLINE: This is a multicenter, phase IIB study followed by a phase III study. Patients are stratified according to institution, age at registration (< 60 years old vs ≥ 60 years old), and presence of liver metastases (yes vs no).

* Phase IIB (step 1): Patients are randomized to 1 of 3 treatment arms.

  * Arm I: Patients receive doxorubicin hydrochloride IV on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive trabectedin IV over 3 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  * Arm III: Patients receive trabectedin IV continuously over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

At the end of step 1, the best regimen of trabectedin will be determined. Patients receiving the non-selected trabectedin regimen ("losing arm") are offered to cross over in order to receive the selected regimen of trabectedin.

* Phase III (step 2): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive trabectedin IV on day 1 using the preferred regimen determined in step 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive doxorubicin hydrochloride IV on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients complete quality of life questionnaire (EORTC QLQ-C30 version 3) at baseline, at 6, 12, 24, and 36 weeks during study, and at the end of study.

Tumor tissue block obtained at diagnosis may be analyzed to identify and validate biomarkers of sensitivity to trabectedin and for tissue microarrays.

After completion of study therapy, patients are followed up at 1 month, every 6 or 12 weeks until disease progression, and every 12 weeks thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed intermediate- or high-grade malignant soft tissue sarcoma

  * Advanced and/or metastatic disease
  * Previously untreated disease
* The following tumor types are not allowed:

  * Well-differentiated liposarcoma
  * Embryonal rhabdomyosarcoma
  * Chondrosarcoma (excluding extraskeletal myxoid chondrosarcoma)
  * Osteosarcoma (excluding extraskeletal osteosarcoma)
  * Ewing tumors/primitive neuroectodermal tumor (PNET)
  * Gastrointestinal stromal tumors (GIST)
  * Dermatofibrosarcoma protuberans
* Must have confirmed disease progression based on investigator's judgment prior to study enrollment
* Measurable disease according to RECIST v 1.1 criteria

  * Tumor lesions situated in a previously irradiated area, or in an area subjected to other loco-regional therapy, are usually not considered measurable unless there has been demonstrated progression in the lesion
* Formalin fixed paraffin embedded tumor blocks or representative hematoxylin/eosin slides (preferably both) available (local histopathological diagnosis will be accepted for trial entry)
* No prior anticancer therapy for this disease

  * No prior anthracycline
  * Non-anthracycline therapy for nonmetastatic disease is acceptable
* No known history of CNS metastases or leptomeningeal tumor spread

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100 x 10^9/L
* Bilirubin normal
* ALT/AST ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN, (if alkaline phosphatase > 2.5 times ULN, hepatic isoenzymes 5-nucleotidase and/or GGT must be within the normal range)
* Albumin > 30 g/L
* Serum creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 30 mL/min
* Creatine phosphokinase (CPK) ≤ 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception (double barrier method for men) 2 weeks prior to, during, and for 3 months (women) or 5 months (men) after completion of study therapy
* LVEF normal by MUGA scan or ECHO
* 12-lead ECG normal (without clinically significant abnormalities)
* None of the following unstable cardiac conditions:

  * Congestive heart failure
  * Angina pectoris
  * Myocardial infarction within the past year
  * Uncontrolled arterial hypertension, defined as BP ≥ 150/100 mm Hg despite optimal medical therapy
  * Clinically significant arrhythmias
* No active or uncontrolled infections or serious illnesses or medical conditions, including a history of any of the following:

  * Chronic alcohol abuse
  * Hepatitis
  * HIV
  * Cirrhosis
* No history of malignancy within the past 5 years, except soft tissue sarcoma, basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, resected incidental prostate cancer (staged pT2 with Gleason score ≤ 6 and postoperative PSA < 0.5 ng/mL)

  * Patients with any history of malignancies who are disease-free for more than 5 years are eligible
* a history of malignancy and disease-free for more than 5 years
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* No concurrent alcohol consumption

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 28 days since prior and no concurrent anticancer therapy including systemic therapy, radiotherapy, or surgery
* At least 28 days since prior and no other concurrent investigational agents
* No concurrent phenytoin, live attenuated vaccines, or yellow fever vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival as assessed by RECIST v 1.1 criteria (phase IIB and phase III)
Safety (phase IIB)

SECONDARY OUTCOMES:
Overall survival (phase III)
Response rate and response duration (phase III)
Safety profile (phase III)
Quality of life (phase III)

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Binh Bui, MD, Study Chair — Institut Bergonié; James E. Butrynski, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (43):
- United States (8):
  - Sarcoma Oncology Center, Santa Monica, California
  - Stanford Hospital and Clinics, Stanford, California
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Dana Farber Institute, Boston, Massachusetts
  - Massachussets General Hospital, Boston, Massachusetts
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Pennsylvania Oncology Hematology Associates, Incorporated - Philadelphia, Philadelphia, Pennsylvania
- Medical University Vienna, Vienna, Austria
- Belgium (3):
  - HôPITAUX UNIVERSITAIRES BORDET-ERASME - INSTITUT JULES BORDET, Brussels
  - Cliniques Universitaires St. Luc, Brussels
  - U.Z. Gasthuisberg, Leuven
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital - University Copenhagen, Herlev
- France (8):
  - Institut Bergonie, Bordeaux
  - Centre Georges-Francois-Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - ASSISTANCE PUBLIQUE - HôPITAUX DE MARSEILLE - HôPITAL DE LA TIMONE, Marseille
  - Institut de Cancerologie de L'Ouest (Ico) - Centre Rene Gauducheau, Nantes - Saint Herblain
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaets-Krankenhaus Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsmedizin Mannheim, Mannheim
  - Klinikum Grosshadern Ludwig-Maximilians Univ. Muenchen, München
- Military Hospital - State Health Centre, Budapest, Hungary
- Netherlands (5):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Erasmus Mc - Daniel Den Hoed Cancer Center, Rotterdam
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- National Cancer Institute, Bratislava, Slovakia
- Spain (2):
  - Hospital General Vall D'Hebron, Barcelona
  - Hospital Universitario San Carlos, Madrid
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (3):
  - Nhs Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre, Glasgow
  - Christie Nhs Foundation Trust, Manchester
  - Nottingham University Hospitals Nhs Trust - City Hospital Campus, Nottingham